CLINICAL TRIAL: NCT07077460
Title: Innovative Hand Rehabilitation System With Synchronized Contralateral Haptic Feedback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Chair Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 113-162
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Healthy Elderly
Keywords: Functional near infrared spectroscopy; Parameters of digit force independence; Mirror Visual Feedback; Hand Training System; Hand Dexterity; Synchronized contralateral haptic feedback

STUDY DESIGN:
Intervention Model Description: Subjects would use their dominant hand to operate the hand training system (Tipr), and according to the game instructions prompted by the tablet screen, slowly press the corresponding finger to the evaluation system to reach the target force value. At the same time, the subjects were instructed to place their non-dominant hand behind the mirror device and place it on another hand training system (Tipr). When the dominant hand starts to execute the game instructions, the force exerted by the fingertips will be presented on the tablet in the form of a game task screen. At the same time, a mirror or other device that can provide a mirror will be used to project the mirrored game screen to the developing device on non-dominant hand side. At the same time, subjects would get the feedback from only mirror visual feedback or both mirror visual feedback and Graded-Pressure Haptic feedback device or no other feedback, respectively for each group, during performing the force control training.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror Visual Feedback Group (Active Comparator): All the subjects were asked to use their dominant hands to operate the hand training system (TIPr) and place their non-dominant hands behind the mirror on the other hand training system (TIPr). According to the game instructions shown on the tablet screen, they should slowly press the evaluation system with the corresponding fingers to reach the target force value. When the dominant hand started to cooperate with the game instructions, the force exerted by the fingertips will be presented on the tablet, and the mirror would show the mirrored (reflected) image of force output level. The subjects were instructed to keep their eyes contacts on the reflected image from the mirror and simultaneously "imagine" that the non-dominant hand performing the same task as the dominant hand. Subjects was instructed not to move their non-dominant hand voluntarily.
  Interventions: Device: TIPr; Device: Mirror Visual Feedback Device
- Non-Mirror Visual Feedback Group (Active Comparator): All the subjects were asked to use their dominant hands to operate the hand training system (TIPr) and place their non-dominant hands behind the mirror on the other hand training system. According to the game instructions shown on the tablet screen, they should slowly press the evaluation system with the corresponding fingers to reach the target force value. When the dominant hand starts to cooperate with the game instructions, the force exerted by the fingertips will be presented on the tablet. Different from MVF group, the mirror would be covered. The subjects were instructed to keep their eyes contact on the tablet and imagine the non-dominant hand performing the same task as the dominant hand without mirror visual feedback. Subjects was instructed not to move their non-dominant hand voluntarily.
  Interventions: Device: TIPr; Device: Mirror Visual Feedback Device(Blocked mirror)
- Output-Dependent Cutaneous Pressure Tactile plus Mirror Visual Feedback Group (Experimental): All the subjects were asked to use their dominant hands to operate the hand training system (TIPr) and place their non-dominant hands behind the mirror on the other hand training system (TIPr). Moreover, graded cutaneous pressure feedback, delivered via a novel Graded-Pressure Haptic Device would be applied on non-dominant fingers. When the dominant hand started to play the game, the force exerted by the fingertips will be presented on the tablet, and the mirror would show the mirrored image of force output level. Subjects were instructed to keep their eyes contacts on the mirrored-image and simultaneously "imagine" that the non-dominant hand performing the same task as the dominant hand. At the same time, subjects would additionally received force pulses on the non-dominant fingertip in synchrony with the TiPR game's force output (matched amplitude) to add tactile feedback. Subjects was instructed not to move their non-dominant hand voluntarily.
  Interventions: Device: TIPr; Device: Mirror Visual Feedback Device; Device: Graded-Pressure Haptic Device (Passive press-feedback cushion)

INTERVENTIONS:
Device: TIPr — TIPr is a second-generation device, which is originated from Pressing Evaluation and Training System (PETs), developed by NCKU Motion Analysis Lab. This 2nd generation device is a home-based training device, which equipped with single-axis force sensors and displayed visual feedback through a tablet advantages.
Device: Mirror Visual Feedback Device — A box with two compartments through a partition with two mirrors installed on each side, which is applied in Mirror therapy.
  Arms: Mirror Visual Feedback Group; Output-Dependent Cutaneous Pressure Tactile plus Mirror Visual Feedback Group
Device: Mirror Visual Feedback Device(Blocked mirror) — Different from Mirror Visual Feedback Device in MVF group, the mirror was blocked by black curtain or paperboard.
  Arms: Non-Mirror Visual Feedback Group
Device: Graded-Pressure Haptic Device (Passive press-feedback cushion) — A passive press-feedback cushion (Graded-Pressure Haptic Device) would deliver force pulses to the subjects' non-dominant fingertips in synchrony with the TiPR game's force output (matched amplitude)
  Arms: Output-Dependent Cutaneous Pressure Tactile plus Mirror Visual Feedback Group

SUMMARY:
Previous studies have found that graded motor imagery (GMI) training can provide continuous activation of the cerebral cortex compared to traditional rehabilitation therapy. One of the steps in this strategy, mirror therapy, has also been widely used in the clinical treatment of hemiplegic patients. Also, comparing with traditional rehabilitation treatments, mirror therapy can continuously provide cortical activation. Besides, several studies indicated that game-based interventions contribute to brain activation in the elderly due to their interest can improve users' motivation in the training program execution. In addition, force control training has positive effects on hand dexterity, and specific doses of motor control training not only improve motor function but also have positive effects on brain function.

Currently, hand function training primarily focuses on range of motion, strength, and hand function, although there is comparatively less emphasis on enhancing both force control and brain function. Moreover, studies related to mirror therapy has primarily focused on the execution of functional movements, but has not explored whether hand strength control training can achieve the same training effects on the affected or non-dominant side through the concept of mirror therapy. Furthermore, the effects of combining a hand strength control system with a synchronous contralateral clip-on force feedback device on brain activation and hand function have not yet been studied. Therefore, this study aimed to investigate the effects of integration a finger force control training system with synchronous contralateral force feedback and mirror visual feedback device on brain activation and hand function, aiming to develop a clinically applicable hand rehabilitation system. Additionally, visual feedback from force control training in our study is through the hints displayed virtually on the game interface of the tablet, which were represented as the height of the targets, not as typical as actual movement-based mirror therapy or task-based mirror therapy.

Therefore, the purpose of the study is to understand the differences among training effects of integrating Graded-Pressure Haptic Device-TiPR closed-loop system and MVF; MVF and force control training, as well as isolated force control training, and to explore the training effects on hand strength, hand function and brain activation.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 20-80 years old
* Without past medical history of musculoskeletal or neurological disorders that would affect muscle control ability or cause sensory abnormalities
* Normal cognitive function to understand and follow the instructions
* Able to understand Chinese, English, or Taiwanese language

Exclusion Criteria:

* With a history of hand-related surgeries
* With a history of neuromuscular diseases or degenerative arthritis
* With a history of brain injury
* With a history of taking psychiatric medications
* Unable to understand instructions, or have cognitive impairments
* With a history of physical disabilities (Loss of body parts) or taking relevant medications, including heart disease, peripheral arterial disease, respiratory system diseases, dialysis, unresolved upper extremity injury, or highly addicted to smoking or alcohol

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-10-22 (Estimated); Study Completion 2025-10-22 (Estimated)

PRIMARY OUTCOMES:
Hand Strength | Before and after intervention(test time:15 minutes)
  Handgrip strength and pinch strength was measured respectively. JAMAR Grip Hand Dynamometer and JAMAR Hydraulic Pinch Gauge were used for the apparatus for force measurement. Pinch strength was divided into lateral pinch, tip pinch and tripod pinch. Each test will test for three times and get the average results.
Purdue Pegboard Test (PPT) | Before and after intervention(total test time for all subtest: 10 minutes)
  Assess the manual dexterity and coordination for one and both hands, including one hand, two hand and assembly subtest. ( Test for dominant hand and non-dominant hand). Each subtest test for three times.
Minnesota Manual Dexterity Test (MMDT) | Before and after intervention(total test time for all subtests:25 minutes)
  Assess the eye-hand coordination ability and manual dexterity. MMDT was divided into: Turning, Placing, One hand Turning and Placing, Two hand Turning and Placing, Displacing.
Digit Independence (EN value) | Before and after intervention(test time:40 seconds for each digits)
  The force independence of each digit is collected from the data during force tracking test in evaluation session. The parameter of force independence is an index of five digits overall enslaving presented as EN value. Dominant hand and non-dominant hand need to be evaluated.
Force control ability | Before and after intervention(test time: 40 seconds for each digits)
  Subjects will be asked to track the target force and presses task digit to fit the target line as accurately as possible. Dominant hand and non-dominant hand need to be evaluated.
Oxygenated hemoglobin (HbO) | Before and after intervention(test time:40 minutes)
  The Oxygenated hemoglobin (HbO) was measured while the participants play the game under both conditions

SECONDARY OUTCOMES:
Maximum voluntary isometric contraction (MVIC) | Every time before the initiation of game(test time:1 seconds for each digit)
  Maximum voluntary isometric contraction of each digit is measured for training reference

CONTACTS AND LOCATIONS:
Overall Officials: Fong-Chin Su, PHD, Principal Investigator — Chair Professor
Locations (1):
- National Cheng Kung University, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim J, Muller KR, Chung YG, Chung SC, Park JY, Bulthoff HH, Kim SP. Distributed functions of detection and discrimination of vibrotactile stimuli in the hierarchical human somatosensory system. Front Hum Neurosci. 2015 Jan 21;8:1070. doi: 10.3389/fnhum.2014.01070. eCollection 2014. PMID 25653609
- [Background] Mendez-Balbuena I, Manjarrez E, Schulte-Monting J, Huethe F, Tapia JA, Hepp-Reymond MC, Kristeva R. Improved sensorimotor performance via stochastic resonance. J Neurosci. 2012 Sep 5;32(36):12612-8. doi: 10.1523/JNEUROSCI.0680-12.2012. PMID 22956850
- [Background] Kim MY, Kwon H, Yang TH, Kim K. Vibration Alert to the Brain: Evoked and Induced MEG Responses to High-Frequency Vibrotactile Stimuli on the Index Finger of Dominant and Non-dominant Hand. Front Hum Neurosci. 2020 Nov 5;14:576082. doi: 10.3389/fnhum.2020.576082. eCollection 2020. PMID 33250728
- [Background] Demain S, Metcalf CD, Merrett GV, Zheng D, Cunningham S. A narrative review on haptic devices: relating the physiology and psychophysical properties of the hand to devices for rehabilitation in central nervous system disorders. Disabil Rehabil Assist Technol. 2013 May;8(3):181-9. doi: 10.3109/17483107.2012.697532. Epub 2012 Jul 16. PMID 22794937
- [Background] Pacheco-Barrios K, Ortega-Marquez J, Fregni F. Haptic Technology: Exploring Its Underexplored Clinical Applications-A Systematic Review. Biomedicines. 2024 Dec 10;12(12):2802. doi: 10.3390/biomedicines12122802. PMID 39767709
- [Background] Dickmann T, Wilhelm NJ, Glowalla C, Haddadin S, van der Smagt P, Burgkart R. An Adaptive Mechatronic Exoskeleton for Force-Controlled Finger Rehabilitation. Front Robot AI. 2021 Sep 30;8:716451. doi: 10.3389/frobt.2021.716451. eCollection 2021. PMID 34660703
- [Background] Sengupta P, Lakshminarayanan K. Motor imagery of finger movements: Effects on cortical and muscle activities. Behav Brain Res. 2024 Aug 5;471:115100. doi: 10.1016/j.bbr.2024.115100. Epub 2024 Jun 7. PMID 38852744
- [Background] Dodakian L, Campbell Stewart J, Cramer SC. Motor imagery during movement activates the brain more than movement alone after stroke: a pilot study. J Rehabil Med. 2014 Oct;46(9):843-8. doi: 10.2340/16501977-1844. PMID 25182189
- [Background] Hsu HY, Chen PT, Kuan TS, Yang HC, Shieh SJ, Kuo LC. A Touch-Observation and Task-Based Mirror Therapy Protocol to Improve Sensorimotor Control and Functional Capability of Hands for Patients With Peripheral Nerve Injury. Am J Occup Ther. 2019 Mar/Apr;73(2):7302205020p1-7302205020p10. doi: 10.5014/ajot.2018.027763. PMID 30915963
- [Background] Kara OK, Yardimci BN, Sahin S, Orhan C, Livanelioglu A, Soylu AR. Combined Effects of Mirror Therapy and Exercises on the Upper Extremities in Children with Unilateral Cerebral Palsy: A Randomized Controlled Trial. Dev Neurorehabil. 2020 May;23(4):253-264. doi: 10.1080/17518423.2019.1662853. Epub 2019 Sep 13. PMID 31514564
- [Background] Arya KN. Underlying neural mechanisms of mirror therapy: Implications for motor rehabilitation in stroke. Neurol India. 2016 Jan-Feb;64(1):38-44. doi: 10.4103/0028-3886.173622. PMID 26754990
- [Background] Bello UM, Winser SJ, Chan CCH. Role of kinaesthetic motor imagery in mirror-induced visual illusion as intervention in post-stroke rehabilitation. Rev Neurosci. 2020 Aug 27;31(6):659-674. doi: 10.1515/revneuro-2019-0106. PMID 32229682
- [Background] Ao D, Song R, Tong KY. Sensorimotor control of tracking movements at various speeds for stroke patients as well as age-matched and young healthy subjects. PLoS One. 2015 Jun 1;10(6):e0128328. doi: 10.1371/journal.pone.0128328. eCollection 2015. PMID 26030289
- [Background] Gowda AS, Memon AN, Bidika E, Salib M, Rallabhandi B, Fayyaz H. Investigating the Viability of Motor Imagery as a Physical Rehabilitation Treatment for Patients With Stroke-Induced Motor Cortical Damage. Cureus. 2021 Mar 19;13(3):e14001. doi: 10.7759/cureus.14001. PMID 33884242
- [Background] Choy CS, Fang Q, Neville K, Ding B, Kumar A, Mahmoud SS, Gu X, Fu J, Jelfs B. Virtual reality and motor imagery for early post-stroke rehabilitation. Biomed Eng Online. 2023 Jul 5;22(1):66. doi: 10.1186/s12938-023-01124-9. PMID 37407988
- [Background] Ji EK, Wang HH, Jung SJ, Lee KB, Kim JS, Jo L, Hong BY, Lim SH. Graded motor imagery training as a home exercise program for upper limb motor function in patients with chronic stroke: A randomized controlled trial. Medicine (Baltimore). 2021 Jan 22;100(3):e24351. doi: 10.1097/MD.0000000000024351. PMID 33546067
- [Background] Park C, Son H. Immediate Effects of Fine-Motor Training on Coordination and Dexterity of the Non-Dominant Hand in Healthy Adults: A Randomized Controlled Trial. Behav Sci (Basel). 2022 Nov 12;12(11):446. doi: 10.3390/bs12110446. PMID 36421742
- [Background] Ehrensberger M, Simpson D, Broderick P, Blake C, Horgan F, Hickey P, O'Reilly J, Monaghan K. Unilateral Strength Training and Mirror Therapy in Patients With Chronic Stroke: A Pilot Randomized Trial. Am J Phys Med Rehabil. 2019 Aug;98(8):657-665. doi: 10.1097/PHM.0000000000001162. PMID 31318745
- [Background] Mulder T. Motor imagery and action observation: cognitive tools for rehabilitation. J Neural Transm (Vienna). 2007;114(10):1265-78. doi: 10.1007/s00702-007-0763-z. Epub 2007 Jun 20. PMID 17579805
- [Background] Fukumura K, Sugawara K, Tanabe S, Ushiba J, Tomita Y. Influence of mirror therapy on human motor cortex. Int J Neurosci. 2007 Jul;117(7):1039-48. doi: 10.1080/00207450600936841. PMID 17613113
- [Background] Formica C, De Salvo S, Muscara N, Bonanno L, Arcadi FA, Lo Buono V, Acri G, Quartarone A, Marino S. Applications of Near Infrared Spectroscopy and Mirror Therapy for Upper Limb Rehabilitation in Post-Stroke Patients: A Brain Plasticity Pilot Study. J Clin Med. 2024 Nov 4;13(21):6612. doi: 10.3390/jcm13216612. PMID 39518751
- [Background] Rosipal R, Porubcova N, Barancok P, Cimrova B, Farkas I, Trejo LJ. Effects of mirror-box therapy on modulation of sensorimotor EEG oscillatory rhythms: a single-case longitudinal study. J Neurophysiol. 2019 Feb 1;121(2):620-633. doi: 10.1152/jn.00599.2018. Epub 2018 Dec 12. PMID 30540503
- [Background] Hamzei F, Lappchen CH, Glauche V, Mader I, Rijntjes M, Weiller C. Functional plasticity induced by mirror training: the mirror as the element connecting both hands to one hemisphere. Neurorehabil Neural Repair. 2012 Jun;26(5):484-96. doi: 10.1177/1545968311427917. Epub 2012 Jan 13. PMID 22247501
- [Background] Zammit AR, Robitaille A, Piccinin AM, Muniz-Terrera G, Hofer SM. Associations Between Aging-Related Changes in Grip Strength and Cognitive Function in Older Adults: A Systematic Review. J Gerontol A Biol Sci Med Sci. 2019 Mar 14;74(4):519-527. doi: 10.1093/gerona/gly046. PMID 29528368
- [Background] Marshall B, Wright DJ, Holmes PS, Wood G. Combining Action Observation and Motor Imagery Improves Eye-Hand Coordination during Novel Visuomotor Task Performance. J Mot Behav. 2020;52(3):333-341. doi: 10.1080/00222895.2019.1626337. Epub 2019 Jun 11. PMID 31185831
- [Background] Kitamura M, Kamibayashi K. Changes in corticospinal excitability during motor imagery by physical practice of a force production task: Effect of the rate of force development during practice. Neuropsychologia. 2024 Aug 13;201:108937. doi: 10.1016/j.neuropsychologia.2024.108937. Epub 2024 Jun 10. PMID 38866222
- [Background] Henschke JU, Pakan JMP. Engaging distributed cortical and cerebellar networks through motor execution, observation, and imagery. Front Syst Neurosci. 2023 Apr 11;17:1165307. doi: 10.3389/fnsys.2023.1165307. eCollection 2023. PMID 37114187
- [Background] Jeannerod M. Neural simulation of action: a unifying mechanism for motor cognition. Neuroimage. 2001 Jul;14(1 Pt 2):S103-9. doi: 10.1006/nimg.2001.0832. PMID 11373140
- [Background] Iwanami J, Mutai H, Sagari A, Sato M, Kobayashi M. Relationship between Corticospinal Excitability While Gazing at the Mirror and Motor Imagery Ability. Brain Sci. 2023 Mar 9;13(3):463. doi: 10.3390/brainsci13030463. PMID 36979273
- [Background] Cengiz B, Vuralli D, Zinnuroglu M, Bayer G, Golmohammadzadeh H, Gunendi Z, Turgut AE, Irfanoglu B, Arikan KB. Analysis of mirror neuron system activation during action observation alone and action observation with motor imagery tasks. Exp Brain Res. 2018 Feb;236(2):497-503. doi: 10.1007/s00221-017-5147-5. Epub 2017 Dec 11. PMID 29230518
- [Background] Kang YJ, Ku J, Kim HJ, Park HK. Facilitation of corticospinal excitability according to motor imagery and mirror therapy in healthy subjects and stroke patients. Ann Rehabil Med. 2011 Dec;35(6):747-58. doi: 10.5535/arm.2011.35.6.747. Epub 2011 Dec 30. PMID 22506202
- [Background] Zhang H, Long Z, Ge R, Xu L, Jin Z, Yao L, Liu Y. Motor imagery learning modulates functional connectivity of multiple brain systems in resting state. PLoS One. 2014 Jan 17;9(1):e85489. doi: 10.1371/journal.pone.0085489. eCollection 2014. PMID 24465577
- [Background] Romkema S, Bongers RM, van der Sluis CK. Influence of mirror therapy and motor imagery on intermanual transfer effects in upper-limb prosthesis training of healthy participants: A randomized pre-posttest study. PLoS One. 2018 Oct 9;13(10):e0204839. doi: 10.1371/journal.pone.0204839. eCollection 2018. PMID 30300378
- [Background] Abdullahi A, Wong TWL, Ng SSM. Rehabilitation of Severe Impairment in Motor Function after Stroke: Suggestions for Harnessing the Potentials of Mirror Neurons and the Mentalizing Systems to Stimulate Recovery. Brain Sci. 2022 Sep 28;12(10):1311. doi: 10.3390/brainsci12101311. PMID 36291245
- [Background] Zapparoli L, Mariano M, Paulesu E. How the motor system copes with aging: a quantitative meta-analysis of the effect of aging on motor function control. Commun Biol. 2022 Jan 20;5(1):79. doi: 10.1038/s42003-022-03027-2. PMID 35058549
- [Background] Lee D, Quessy S. Activity in the supplementary motor area related to learning and performance during a sequential visuomotor task. J Neurophysiol. 2003 Feb;89(2):1039-56. doi: 10.1152/jn.00638.2002. PMID 12574479
- [Background] Leo A, Handjaras G, Bianchi M, Marino H, Gabiccini M, Guidi A, Scilingo EP, Pietrini P, Bicchi A, Santello M, Ricciardi E. A synergy-based hand control is encoded in human motor cortical areas. Elife. 2016 Feb 15;5:e13420. doi: 10.7554/eLife.13420. PMID 26880543
- [Background] Ehrsson HH, Fagergren A, Jonsson T, Westling G, Johansson RS, Forssberg H. Cortical activity in precision- versus power-grip tasks: an fMRI study. J Neurophysiol. 2000 Jan;83(1):528-36. doi: 10.1152/jn.2000.83.1.528. PMID 10634893
- [Background] Spraker MB, Corcos DM, Vaillancourt DE. Cortical and subcortical mechanisms for precisely controlled force generation and force relaxation. Cereb Cortex. 2009 Nov;19(11):2640-50. doi: 10.1093/cercor/bhp015. Epub 2009 Mar 2. PMID 19254959
- [Background] Paclet F, Quaine F. Motor control theories improve biomechanical model of the hand for finger pressing tasks. J Biomech. 2012 Apr 30;45(7):1246-51. doi: 10.1016/j.jbiomech.2012.01.038. Epub 2012 Feb 20. PMID 22356843
- [Background] Zhang N, Yuan X, Li Q, Wang Z, Gu X, Zang J, Ge R, Liu H, Fan Z, Bu L. The effects of age on brain cortical activation and functional connectivity during video game-based finger-to-thumb opposition movement: A functional near-infrared spectroscopy study. Neurosci Lett. 2021 Feb 16;746:135668. doi: 10.1016/j.neulet.2021.135668. Epub 2021 Jan 23. PMID 33497717
- [Background] Seol J, Lim N, Nagata K, Okura T. Effects of home-based manual dexterity training on cognitive function among older adults: a randomized controlled trial. Eur Rev Aging Phys Act. 2023 Apr 22;20(1):9. doi: 10.1186/s11556-023-00319-2. PMID 37087432
- [Background] Lin CH, Sung WH, Chiang SL, Lee SC, Lu LH, Wang PC, Wang XM. Influence of aging and visual feedback on the stability of hand grip control in elderly adults. Exp Gerontol. 2019 May;119:74-81. doi: 10.1016/j.exger.2019.01.024. Epub 2019 Jan 26. PMID 30695717
- [Background] Klemm L, Kuehn E, Kalyani A, Schreiber S, Reichert C, Azanon E. Age-related differences in finger interdependence during complex hand movements. J Appl Physiol (1985). 2024 Jul 1;137(1):181-193. doi: 10.1152/japplphysiol.00606.2023. Epub 2024 May 2. PMID 38695353
- [Background] Vieluf S, Godde B, Reuter EM, Voelcker-Rehage C. Age-related differences in finger force control are characterized by reduced force production. Exp Brain Res. 2013 Jan;224(1):107-17. doi: 10.1007/s00221-012-3292-4. Epub 2012 Oct 18. PMID 23076430
- [Background] Kraeutner SN, Rubino C, Ferris JK, Rinat S, Penko L, Chiu L, Greeley B, Jones CB, Larssen BC, Boyd LA. Frontoparietal function and underlying structure reflect capacity for motor skill acquisition during healthy aging. Neurobiol Aging. 2024 Jan;133:78-86. doi: 10.1016/j.neurobiolaging.2023.10.007. Epub 2023 Oct 20. PMID 37918189
- [Background] Kleerekooper I, van Rooij SJH, van den Wildenberg WPM, de Leeuw M, Kahn RS, Vink M. The effect of aging on fronto-striatal reactive and proactive inhibitory control. Neuroimage. 2016 May 15;132:51-58. doi: 10.1016/j.neuroimage.2016.02.031. Epub 2016 Feb 17. PMID 26899783
- [Background] Olafsdottir HB, Zatsiorsky VM, Latash ML. The effects of strength training on finger strength and hand dexterity in healthy elderly individuals. J Appl Physiol (1985). 2008 Oct;105(4):1166-78. doi: 10.1152/japplphysiol.00054.2008. Epub 2008 Aug 7. PMID 18687981
- [Background] Heintz Walters B, Huddleston WE, O'Connor K, Wang J, Hoeger Bement M, Keenan KG. Visual feedback and declines in attention are associated with altered visual strategy during a force-steadiness task in older adults. J Neurophysiol. 2023 Nov 1;130(5):1309-1320. doi: 10.1152/jn.00486.2022. Epub 2023 Oct 25. PMID 37877175
- [Background] Manelis A, Hu H, Satz S. The Relationship Between Reduced Hand Dexterity and Brain Structure Abnormality in Older Adults. Geriatrics (Basel). 2024 Dec 17;9(6):165. doi: 10.3390/geriatrics9060165. PMID 39727824
- [Background] Hesseberg K, Tangen GG, Pripp AH, Bergland A. Associations between Cognition and Hand Function in Older People Diagnosed with Mild Cognitive Impairment or Dementia. Dement Geriatr Cogn Dis Extra. 2020 Dec 15;10(3):195-204. doi: 10.1159/000510382. eCollection 2020 Sep-Dec. PMID 33569075
- [Background] Incel NA, Sezgin M, As I, Cimen OB, Sahin G. The geriatric hand: correlation of hand-muscle function and activity restriction in elderly. Int J Rehabil Res. 2009 Sep;32(3):213-8. doi: 10.1097/MRR.0b013e3283298226. PMID 19293723
- [Background] Mates J, Muller U, Radil T, Poppel E. Temporal integration in sensorimotor synchronization. J Cogn Neurosci. 1994 Fall;6(4):332-40. doi: 10.1162/jocn.1994.6.4.332. PMID 23961729
- [Background] Edin BB, Westling G, Johansson RS. Independent control of human finger-tip forces at individual digits during precision lifting. J Physiol. 1992 May;450:547-64. doi: 10.1113/jphysiol.1992.sp019142. PMID 1432717
- [Background] Ambike SS, Paclet F, Latash ML, Zatsiorsky VM. Grip-force modulation in multi-finger prehension during wrist flexion and extension. Exp Brain Res. 2013 Jun;227(4):509-22. doi: 10.1007/s00221-013-3527-z. Epub 2013 Apr 30. PMID 23625077
- [Background] Guan J, Wade MG. The effect of aging on adaptive eye-hand coordination. J Gerontol B Psychol Sci Soc Sci. 2000 May;55(3):P151-62. doi: 10.1093/geronb/55.3.p151. PMID 11833977
- [Background] Stockel T, Wunsch K, Hughes CML. Age-Related Decline in Anticipatory Motor Planning and Its Relation to Cognitive and Motor Skill Proficiency. Front Aging Neurosci. 2017 Sep 4;9:283. doi: 10.3389/fnagi.2017.00283. eCollection 2017. PMID 28928653
- [Background] Kovalev VA, Kruggel F, von Cramon DY. Gender and age effects in structural brain asymmetry as measured by MRI texture analysis. Neuroimage. 2003 Jul;19(3):895-905. doi: 10.1016/s1053-8119(03)00140-x. PMID 12880818
- [Background] Ueno M, Nakamura Y, Li J, Gu Z, Niehaus J, Maezawa M, Crone SA, Goulding M, Baccei ML, Yoshida Y. Corticospinal Circuits from the Sensory and Motor Cortices Differentially Regulate Skilled Movements through Distinct Spinal Interneurons. Cell Rep. 2018 May 1;23(5):1286-1300.e7. doi: 10.1016/j.celrep.2018.03.137. PMID 29719245
- [Background] Heffner RS, Masterton RB. The role of the corticospinal tract in the evolution of human digital dexterity. Brain Behav Evol. 1983;23(3-4):165-83. doi: 10.1159/000121494. PMID 6667369
- [Background] Rozand V, Senefeld JW, Sundberg CW, Smith AE, Hunter SK. Differential effects of aging and physical activity on corticospinal excitability of upper and lower limb muscles. J Neurophysiol. 2019 Jul 1;122(1):241-250. doi: 10.1152/jn.00077.2019. Epub 2019 May 15. PMID 31091158
- [Background] Blinkouskaya Y, Cacoilo A, Gollamudi T, Jalalian S, Weickenmeier J. Brain aging mechanisms with mechanical manifestations. Mech Ageing Dev. 2021 Dec;200:111575. doi: 10.1016/j.mad.2021.111575. Epub 2021 Oct 1. PMID 34600936
- [Background] Liu X, Tyler LK, Cam-Can, Davis SW, Rowe JB, Tsvetanov KA. Cognition's dependence on functional network integrity with age is conditional on structural network integrity. Neurobiol Aging. 2023 Sep;129:195-208. doi: 10.1016/j.neurobiolaging.2023.06.001. Epub 2023 Jun 6. PMID 37392579
- [Background] Chen Q, Xia Y, Zhuang K, Wu X, Liu G, Qiu J. Decreased inter-hemispheric interactions but increased intra-hemispheric integration during typical aging. Aging (Albany NY). 2019 Nov 21;11(22):10100-10115. doi: 10.18632/aging.102421. Epub 2019 Nov 21. PMID 31761785
- [Background] de Leeuw FE, de Groot JC, Achten E, Oudkerk M, Ramos LM, Heijboer R, Hofman A, Jolles J, van Gijn J, Breteler MM. Prevalence of cerebral white matter lesions in elderly people: a population based magnetic resonance imaging study. The Rotterdam Scan Study. J Neurol Neurosurg Psychiatry. 2001 Jan;70(1):9-14. doi: 10.1136/jnnp.70.1.9. PMID 11118240
- [Background] Seidler RD, Bernard JA, Burutolu TB, Fling BW, Gordon MT, Gwin JT, Kwak Y, Lipps DB. Motor control and aging: links to age-related brain structural, functional, and biochemical effects. Neurosci Biobehav Rev. 2010 Apr;34(5):721-33. doi: 10.1016/j.neubiorev.2009.10.005. Epub 2009 Oct 20. PMID 19850077
- [Background] Morrison JH, Baxter MG. The ageing cortical synapse: hallmarks and implications for cognitive decline. Nat Rev Neurosci. 2012 Mar 7;13(4):240-50. doi: 10.1038/nrn3200. PMID 22395804
- [Background] Navakkode S, Kennedy BK. Neural ageing and synaptic plasticity: prioritizing brain health in healthy longevity. Front Aging Neurosci. 2024 Aug 5;16:1428244. doi: 10.3389/fnagi.2024.1428244. eCollection 2024. PMID 39161341
- [Background] Cleeland C, Pipingas A, Scholey A, White D. Neurochemical changes in the aging brain: A systematic review. Neurosci Biobehav Rev. 2019 Mar;98:306-319. doi: 10.1016/j.neubiorev.2019.01.003. Epub 2019 Jan 6. PMID 30625337
- [Background] Leisman G, Moustafa AA, Shafir T. Thinking, Walking, Talking: Integratory Motor and Cognitive Brain Function. Front Public Health. 2016 May 25;4:94. doi: 10.3389/fpubh.2016.00094. eCollection 2016. PMID 27252937
- [Background] Hunter SK, Pereira HM, Keenan KG. The aging neuromuscular system and motor performance. J Appl Physiol (1985). 2016 Oct 1;121(4):982-995. doi: 10.1152/japplphysiol.00475.2016. Epub 2016 Aug 11. PMID 27516536
- [Background] Ma Y, Fu L, Jia L, Han P, Kang L, Yu H, Chen X, Yu X, Hou L, Wang L, Zhang W, Niu K, Guo Q. Muscle strength rather than muscle mass is associated with osteoporosis in older Chinese adults. J Formos Med Assoc. 2018 Feb;117(2):101-108. doi: 10.1016/j.jfma.2017.03.004. Epub 2017 Apr 13. PMID 28416075
- [Background] Volpi E, Nazemi R, Fujita S. Muscle tissue changes with aging. Curr Opin Clin Nutr Metab Care. 2004 Jul;7(4):405-10. doi: 10.1097/01.mco.0000134362.76653.b2. PMID 15192443
- [Background] Holloszy JO. The biology of aging. Mayo Clin Proc. 2000 Jan;75 Suppl:S3-8; discussion S8-9. PMID 10959208
- [Background] Power GA, Dalton BH, Rice CL. Human neuromuscular structure and function in old age: A brief review. J Sport Health Sci. 2013 Dec;2(4):215-226. doi: 10.1016/j.jshs.2013.07.001. PMID 27011872
- [Background] Kim HW, Lee DG. Resting-State Metabolism of Hand Knob Area on 18F-FDG PET-CT According to Hand Function and Tractography of Corticospinal Tract After Stroke. Ann Rehabil Med. 2017 Apr;41(2):171-177. doi: 10.5535/arm.2017.41.2.171. Epub 2017 Apr 27. PMID 28503448
- [Background] Lee J, Kim HJ. Normal Aging Induces Changes in the Brain and Neurodegeneration Progress: Review of the Structural, Biochemical, Metabolic, Cellular, and Molecular Changes. Front Aging Neurosci. 2022 Jun 30;14:931536. doi: 10.3389/fnagi.2022.931536. eCollection 2022. PMID 35847660
- [Background] Lopez-Otin C, Blasco MA, Partridge L, Serrano M, Kroemer G. Hallmarks of aging: An expanding universe. Cell. 2023 Jan 19;186(2):243-278. doi: 10.1016/j.cell.2022.11.001. Epub 2023 Jan 3. PMID 36599349
- [Background] Zhu L, Fratiglioni L, Guo Z, Aguero-Torres H, Winblad B, Viitanen M. Association of stroke with dementia, cognitive impairment, and functional disability in the very old: a population-based study. Stroke. 1998 Oct;29(10):2094-9. doi: 10.1161/01.str.29.10.2094. PMID 9756588
- [Background] Zhang J, Sun Y, Li A. The prevalence of disability in older adults with multimorbidity: a meta-analysis. Aging Clin Exp Res. 2024 Sep 10;36(1):186. doi: 10.1007/s40520-024-02835-2. PMID 39254880
- [Background] Wolff JL, Starfield B, Anderson G. Prevalence, expenditures, and complications of multiple chronic conditions in the elderly. Arch Intern Med. 2002 Nov 11;162(20):2269-76. doi: 10.1001/archinte.162.20.2269. PMID 12418941
- [Background] Harman D. Aging: overview. Ann N Y Acad Sci. 2001 Apr;928:1-21. doi: 10.1111/j.1749-6632.2001.tb05631.x. PMID 11795501
- [Background] Ranganathan VK, Siemionow V, Sahgal V, Yue GH. Effects of aging on hand function. J Am Geriatr Soc. 2001 Nov;49(11):1478-84. doi: 10.1046/j.1532-5415.2001.4911240.x. PMID 11890586